CLINICAL TRIAL: NCT06723236
Title: A Phase 1, First-in-Human, Open Label, Dose Escalation and Cohort Expansion Study of MGC028 in Participants With Advanced Solid Tumors
Brief Title: A Study of MGC028 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGC028-01
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors; NSCLC Adenocarcinoma; Cholangiocarcinoma; Pancreatic Carcinoma; Colorectal Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): Dose level 1 of MGC028, IV
  Interventions: Biological: MGC028
- Cohort 2 (Experimental): Dose level 2 of MGC028, IV
  Interventions: Biological: MGC028
- Cohort 3 (Experimental): Dose level 3 of MGC028, IV
  Interventions: Biological: MGC028
- Cohort 4 (Experimental): Dose level 4 of MGC028, IV
  Interventions: Biological: MGC028
- Cohort 5 (Experimental): Dose level 5 of MGC028, IV
  Interventions: Biological: MGC028
- Cohort 6 (Experimental): Dose level 6 of MGC028, IV
  Interventions: Biological: MGC028
- Expansion Cohort 1 (Experimental): MTD or MAD of MGC028, IV
  Interventions: Biological: MGC028
- Expansion Cohort 2 (Experimental): MTD or MAD of MGC028, IV
  Interventions: Biological: MGC028
- Expansion Cohort 3 (Experimental): MTD or MAD of MGC028, IV
  Interventions: Biological: MGC028

INTERVENTIONS:
Biological: MGC028 — MGC028 is an antibody-drug conjugate targeted against ADAM9.

SUMMARY:
The goal of this clinical trial is to characterize the safety, tolerability, dose-limiting toxicities (DLT), and maximum tolerated dose (MTD) or maximum administered dose of MGC028 (if no MTD is defined). The study will enroll adult participants with relapsed or refractory, unresectable, locally advanced of metastatic solid tumors known to express ADAM9.

The main question the study aims to answer is:

* What types of side effects will participants experience when receiving MGC028?
* Can MGC028 cause cancer to shrink, remain stable, or able to control disease progression of participants with advanced solid tumors?

Participants will

* Undergo screening procedures to determine eligibility
* Receive study treatments initially every 3 weeks.
* Have blood samples taken for routine and research tests
* Have other examinations to check heart and lung function, and general health status
* Be asked about any side effects that may be happening or other medications you are taking. The study doctor will provide treatment for side effects, if necessary.
* Have the study doctor assess your tumor status at regular intervals to determine how you are responding to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants in dose escalation or supplemental cohorts must have histologically proven unresectable, locally advanced or metastatic solid tumor limited to one of the following types: NSCLC adenocarcinoma, cholangiocarcinoma, colorectal carcinoma (CRC), or pancreatic carcinoma that is refractory to standard therapy, or for which standard therapy does not exist, has proven to be intolerable, or has been refused by the participant.
* Participants in expansion cohorts must have either

  * NSCLC adenocarcinoma with

    * progression on or following anti-PD-1/PD-L1 inhibitor, unless contraindicated
    * progression on or following therapy for actionable mutations (e.g. EGFR or ALK mutations), if present
    * no more than 2 prior lines of cytotoxic chemotherapy for advanced or metastatic disease.
  * Pancreatic cancer

    * following at least 1 systemic therapy
    * no more than 2 prior lines of cytotoxic therapy for advanced or metastatic disease.
  * Colorectal adenocarcinoma with

    * Progression during or following standard therapy with a fluoropyrimidine-based chemotherapy, oxaliplatin and irinotecan unless contraindicated, refused or unavailable
    * Progression after prior targeted treatment for CRC with actionable mutations such as EGFR, KRAS, BRAF and MSI- H/dMMR, if present.
    * No more that 2 lines of cytotoxic chemotherapy for advanced or metastatic disease
    * No more than 4 lines of systemic regimens for advanced or metastatic disease
* Participants must have at least one lesion that meets the definition of measurable disease by RECIST v1.1.
* Participants must have an available archival or formalin-fixed paraffin-embedded tumor tissue or be willing to undergo a biopsy procedure to obtain a fresh tumor sample.
* Participants have acceptable physical condition and laboratory values.
* Participants of childbearing potential must agree to use highly effective methods of birth control.
* Participants must not be pregnant, planning to be pregnant, or breastfeeding.

Exclusion Criteria:

* Any underlying medical or psychiatric condition impairing participant's ability to receive, tolerate, or comply with the planned treatment or study procedures.
* Active brain metastases or leptomeningeal metastases.
* Prior stem cell, tissue, or solid organ transplant.
* Another malignancy that required treatment within the past 2 years, with the exception of those with a negligible risk of metastasis or death such as adequately treated non-melanomatous skin cancer, localized prostate cancer (Gleason Score < 6), or carcinoma in situ.
* Active viral, bacterial, or fungal infection
* Prior treatment with ADAM9 targeted agent for cancer.
* Prior treatment with major surgery, mediastinal or lung radiation, vaccination with live virus vaccines, systemic cancer treatment, chimeric antigen receptor (CAR)-T cell therapy, or experimental treatment within 4 weeks of the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number and Types of Adverse Events (AEs) in Participants Receiving MGC028 | Throughout the study treatment and safety follow up period, up to 25 months
  Types of AEs include Serious Adverse Events (SAEs), and AEs Leading to Treatment Delay or Discontinuation or Dose Reduction, dose limiting toxicities, and AEs of Special Interest. Observation of side effects determines the highest safe dose for further study

SECONDARY OUTCOMES:
Mean maximum concentration of MGC028 antibody | Through Cycle 6 of the study, approximately 18 weeks
  Measurement of the highest concentration of MGC028 conjugated and total antibody in the bloodstream.
Mean Area Under the Concentration Time Curve of MGC028 antibody | Through Cycle 6 of the study, approximately 18 weeks
  Measurement of the total exposure of MGC028 conjugated and total antibody in the bloodstream.
Number of Participants Who Develop Anti-Drug Antibodies to MGC028 | Throughout the study treatment period, up to 2 years
Objective Response Rate (ORR) | Throughout the study and follow up period, up to 2.5 years.
  The ORR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is estimated as the proportion of participants in the Response Evaluable Population who achieve Best Overall Response of Complete Response or Partial Response.
Median Duration of Response | Throughout the study and follow up period, up to 2.5 years.
  DoR is defined as the time from the date of initial response (CR or PR) to the date of first documented progression or death from any cause, whichever occurs first.
Mean maximum concentration of MGC028 free payload | Through Cycle 6 of the study, approximately 18 weeks
  Measurement of the highest concentration of MGC028 free payload in the bloodstream.
Mean Area Under the Concentration Time Curve Total exposure of MGC028 payload | Through Cycle 6 of the study, approximately 18 weeks
  Measurement of the total exposure of MGC028 free payload in the bloodstream
Change from baseline in the level of ADAM9 expression in tumor specimens, using immunohistochemistry | Baseline and approximately 28 days after the first dose of MGC028.

CONTACTS AND LOCATIONS:
Overall Officials: Pepi Pencheva, M.D., Study Director — MacroGenics
Locations (6):
- United States (6):
  - UCSF - Helen Diller Family Cancer Center, San Francisco, California
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - South Texas Accelerated Research Therapeutics (START) San Antonio, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START) Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scribner JA, Brown JG, Son T, Jin L, McKenzie C, Nam V, Bush C, Quinonez D, Ford D, Tamura J, Gorlatov S, Summers A, Hav M, Li H, Sharma NK, Zhang X, Diedrich G, Butler S, Bonvini E, Loo D. Preclinical development of MGC028, an ADAM9-targeted, glycan-linked, exatecan-based antibody-drug conjugate for the treatment of solid cancers. Mol Cancer Ther. 2025 Oct 30. doi: 10.1158/1535-7163.MCT-25-0461. Online ahead of print. PMID 41166694